CLINICAL TRIAL: NCT01594502
Title: R01 CA155301: Validation of Digital Morphometry for Cancer Risk in Benign Prostate Biopsies
Brief Title: Validation of Digital Morphometry for Cancer Risk in Benign Prostate Biopsies
Status: Completed | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Peter Gann, Professor and Director, Division of Pathology Research, University of Illinois at Chicago
Other Study IDs: 2010-0670; R01CA155301 (NIH)
Record Dates: First submitted 2012-04-17; First posted 2012-05-09 (Estimated); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; dutasteride
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dutasteride

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Biopsy tissue (Year 2 and Year 4) already collected in REDUCE trial
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Dutasteride Year 2 PCa: Subject assigned to dutasteride, prostate cancer found on Year 2 biopsy.
  Interventions: Drug: Dutasteride
- Placebo Year 2 no PCa, Year 4 PCa: Subject assigned to placebo, no prostate cancer found on Year 2 biopsy, but prostate cancer found on Year 4 biopsy.
  Interventions: Drug: Placebo
- Dutasteride Year 2 no PCa, Year 4 PCa: Subject assigned to dutasteride, no prostate cancer found on Year 2 biopsy, but prostate cancer found on Year 4 biopsy.
  Interventions: Drug: Dutasteride
- Placebo, Year 2 and 4 no PCa: Subject assigned to placebo, no prostate cancer found on Year 2 or Year 4 biopsy.
  Interventions: Drug: Placebo
- Dutasteride, Year 2 and 4 no PCa: Subject assigned to dutasteride, no prostate cancer found on Year 2 or Year 4 biopsy.
  Interventions: Drug: Dutasteride
- Placebo, Year 2 PCa: Subject assigned to placebo, prostate cancer found on Year 2 biopsy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dutasteride — 0.5 mg daily
  Groups: Dutasteride Year 2 PCa; Dutasteride Year 2 no PCa, Year 4 PCa; Dutasteride, Year 2 and 4 no PCa
Drug: Placebo — Placebo Comparator
  Groups: Placebo Year 2 no PCa, Year 4 PCa; Placebo, Year 2 PCa; Placebo, Year 2 and 4 no PCa

SUMMARY:
The goal of this study is to apply cutting-edge imaging approaches, incorporating machine-learning for pattern recognition and multispectral analysis, to the development and validation of intermediate endpoint biomarkers in benign tissue that characterize the response to 5α-reductase inhibitor chemoprevention as well as the risk of prostate cancer among men with negative biopsies.

ELIGIBILITY:
Inclusion Criteria:

* completed REDUCE trial (Year 4 exit biopsy with blocks and HE slides available; i.e., U.S. participants only)
* compliant with assigned treatment based on either: (dutasteride group) at least 3 post-baseline serum DHT levels ≥ 50% lower than baseline, or (placebo group) at least 3 post-baseline serum DHT levels with none showing ≥ 50% decrease from baseline

Exclusion Criteria:

* N/A

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Probability Sample
Sampling Method: Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2011-09; Primary Completion 2015-11 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Effects of dutasteride (vs. placebo) using multi-feature scores derived from digital image analysis on both nuclear and architectural features in benign prostate tissue. | Year 4

SECONDARY OUTCOMES:
Multivariable treatment-response score between subjects who develop PCa while on dutasteride and those who do not. | Year 4
Magnitude of association between nuclear phenotype in benign biopsies, and subsequent risk of PCa in untreated men at elevated risk. | Year 4

CONTACTS AND LOCATIONS:
Overall Officials: Peter H Gann, MD, ScD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States